CLINICAL TRIAL: NCT07302984
Title: Mind-body Skills Groups for the Treatment of War-Related Trauma in Adolescents in Gaza: A Randomized Controlled Study
Brief Title: Mind-body Skills Groups for War-Related Trauma in Adolescents in Gaza
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: Americares (Other)
Responsible Party: Principal Investigator, Jamil Abdel Atti, Country Director, The Center for Mind-Body Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GT-CMBM-003
Record Dates: First submitted 2025-12-07; First posted 2025-12-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: meditation; guided imagery; PTSD; mind-body medicine; adolescents
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-Body Skills Groups (Experimental)
  Interventions: Behavioral: Mind-Body Skills Groups
- Wait List Control (No Intervention)

INTERVENTIONS:
Behavioral: Mind-Body Skills Groups — Small group intervention consisting of guided imagery, slow deep breathing, autogenic training, drawings, and active techniques.
  Arms: Mind-Body Skills Groups

SUMMARY:
The goal of this clinical trial is to learn if mind-body skills groups can reduce posttraumatic stress disorder and emotional and behavioral problems in war-traumatized adolescents in Gaza.

The main questions it aims to answer are:

* Do mind-body skills groups reduce posttraumatic stress disorder symptoms in war-traumatized adolescents in Gaza?
* Do mind-body skills groups reduce emotional and behavioral problems in war-traumatized adolescents in Gaza?

Researchers will compare the results of adolescents who do not attend mind-body skills groups to adolescents who attend mind-body skills groups see if those who attend groups have less posttraumatic stress disorder symptoms and emotional and behavioral problems.

Participants will:

* Be screened to determine whether they qualify to be in the study
* If they qualify, they will attend 5 mind-body skills group sessions (if they are not in the control group)
* Fill out research packets before the first session, after the last session, and at 2-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* being 11-17 years old and living in Gaza
* having experienced a political violence or war-related criterion A stressor
* meeting the American Psychiatric Association (APA) Diagnostic and Statistical Manual-(DSM-5-TR) criteria for PTSD according to the screening cut-off score on the Child PTSD Symptom Scale-5 (CPSS-5).

Exclusion Criteria:

* former psychotherapy or medication to treat mental disorders
* having significant cognitive impairment.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Child Post-Traumatic Stress Disorder Symptom Scale - 5 | Before first group session, 2 weeks, 2 months
  Self-report Post-Traumatic Stress Disorder symptom scale with scores from 0 to 80. Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Youth Pediatric Symptom Checklist-17 | Before first group session, 2 weeks, 2 months
  Assessment of Psychosocial Functioning with score range 0 - 34. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Julie K. Staples, PhD, Study Director — The Center for Mind-Body Medicine
Locations (1):
- The Center for Mind-Body Medicine, Deir al-Balah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual patient data
Time Frame: Beginning upon publication of the results
Access Criteria: Anyone may access the de-identified individual patient data through supplemental material published by the journal

REFERENCES:
- [Background] Staples JK, Abdel Atti JA, Gordon JS. Mind-body skills groups for posttraumatic stress disorder and depression symptoms in Palestinian children and adolescents in Gaza. Int J Stress Manag. 2011; 18(3): 246-262. doi:/10.1037/trm0000081
- See also: The organization's website — https://cmbm.org/